CLINICAL TRIAL: NCT00832520
Title: INST 0816: Phase II Study of Remeron for Cancer Patients Losing More Than 10% of Their Body Weight
Brief Title: Phase II Study of Remeron for Cancer Patients Losing More Than 10% of Their Body Weight
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INST 0816
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer; weight loss; Remeron; body weight
MeSH Terms: conditions — Weight Loss; Body Weight | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Remeron (Mirtazapine) (Experimental): Mirtazapine 15 mg orally at bed time for 8 weeks
  Interventions: Drug: Remeron (mirtazapine)

INTERVENTIONS:
Drug: Remeron (mirtazapine) — Mirtazapine 15 mg orally at bed time. Patients with a creatinine clearance < 50% or a bilirubin or transaminases > twice the upper limit of normal will take a 7.5 mg dose.
  * Drug Administration: Drug will be administered orally, every day for a period of 8 weeks
  * Dose modifications: None
  Other Names: mirtazapine

SUMMARY:
The purpose of this study is to find out if remeron, also called mirtazapine, can help you prevent weight loss while on treatment for your cancer. Remeron is currently used to treat depression and has not been approved by the Food and Drug Administration for use to treat weight loss.

DETAILED DESCRIPTION:
Weight loss in cancer patients can be the result of inadequate intake or absorption of nutrients and/or tumor-induced weight loss due to metabolic changes the tumor is creating in the body (1). Inadequate intake resulting in a starvation state can simply be the result of eating less due to depression, nausea/vomiting, feelings of fullness, and taste changes (2). Though not intentional the weight loss caused by these symptoms can be explained and reversed by increasing intake of nutrients. Unintentional weight loss induced by the tumor can be caused by multiple physiological factors that increase the catabolism of muscle and fat and increased nutrient intake alone may not reverse the weight loss. Unintentional weight loss can predict a poor prognosis in cancer patients which is most likely due to decreased doses of treatment (3-5).

Usual care for weight loss in cancer patients varies among practitioners and can include nutrition counseling by a registered dietitian or by the practitioner themselves. Treatment can vary from counseling patients to increase intake of nutrient dense foods to prescribing medications in order to improve appetite or mood, to decrease feelings of fullness, or to control nausea/vomiting, etc. (6). However, these interventions do not always work. For varied reasons not all patients are able to improve their oral intake of food items and in patients with tumor induced weight loss increased oral intake does not improve the metabolic changes.

Anti-depressant medications have weight related side effects (7-9). Mirtazapine has been shown to have side effects of increased appetite and increased weight in cancer subjects studied for use with depression and nausea. (10-13). These results appeared to range from changes in appetite to changes seen in metabolic processes such as changes in the cytokine system to reduce inflammation seen in cachectic patients. Therefore, using mirtazapine in cancer patients even without depression may help to stop unwanted weight loss and increase survival by allowing patient to complete prescribed treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older, with advanced cancer are eligible.
2. Patients must have lost 10% in the last 6 months
3. Patients must have a life expectancy of at least 12 weeks.
4. Patients must have a Zubrod performance status of 0-3.
5. Patients must sign an informed consent.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded from this study.
2. Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
3. Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
4. Patients with head and neck cancers and GI cancers who have functional problems that limits food intake or absorption of nutrients such as partial or complete bowel obstructions, and patients with skin cancers (except melanoma) are not eligible
5. Patients who lost weight on a voluntary diet.
6. Patients who are already taking an appetite stimulant or other anti-depressant, except for SSRI taken in the morning.
7. Patients who had surgery in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - Universtiy of New Mexico - Cancer Center, Albuquerque, New Mexico

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was low (13 of a target 59) which rendered planned statistical analyses impossible. The recruitment period spanned 07Apr2009 through 14Jul2010. All were recruited through the UNM Cancer Center medical clinic.
Period: Overall Study
Arm/Group | Remeron (Mirtazapine)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Remeron (Mirtazapine)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: 8 weeks
Population: There will be no publication, as this study was terminated after the original PI left employment with the institution, and because enrollment was low (13 of a target 59) which rendered planned statistical analyses impossible.
Arm/Group | Remeron (Mirtazapine)
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine if the Quality of Life Improves After Starting Mirtazapine
Time Frame: 8 weeks
Population: as for outcome 1
Arm/Group | Remeron (Mirtazapine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Regular investigator assessment, regular laboratory testing, and self-reporting by subjects.
Arm/Group | Remeron (Mirtazapine)
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remeron (Mirtazapine) (N=13)
Agitation (Psychiatric disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to no subjects analyzed.There will be no publication, as this study was terminated after the original PI left employment with the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No